CLINICAL TRIAL: NCT07194850
Title: A Multicenter, Randomized, Double-blinded, Parallel-Arm, Placebo-Controlled, Pharmacokinetic and Pharmacodynamic Study Followed by an Open-Label Arm to Evaluate Efgartigimod IV in Pediatric Participants From 12 Years to Less Than 18 Years of Age With Chronic ITP
Brief Title: A Study of Efgartigimod IV in Participants From 12 Years to Less Than 18 Years of Age With Chronic Immune Thrombocytopenia (ITP)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-2409; 2025-521055-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-19; First posted 2025-09-26 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Immune Thrombocytopenia (ITP); ITP - Immune Thrombocytopenia; ITP; Immune Thrombocytopenic Purpura; Immune Thrombocytopenic Purpura ( ITP ); Idiopathic Thrombocytopenic Purpura; Idiopathic Thrombocytopenic Purpura (ITP)
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efgartigimod IV (Experimental): Participants receiving efgartigimod IV during the double-blinded treatment period and the open-label treatment period(s)
  Interventions: Biological: Efgartigimod IV
- Placebo IV (Placebo Comparator): Participants receiving placebo IV during the double-blinded treatment period and receiving efgartigimod IV during the open-label treatment period(s)
  Interventions: Biological: Efgartigimod IV; Other: Placebo IV

INTERVENTIONS:
Biological: Efgartigimod IV — Intravenous infusion of efgartigimod
Other: Placebo IV — Intravenous infusion of placebo
  Arms: Placebo IV

SUMMARY:
The main purpose of this study is to confirm the correct dose of efgartigimod IV for treating patients aged 12 to younger than 18 years with chronic immune thrombocytopenia (ITP).

The study consists of a double-blinded treatment period (DBTP) in which the participants will be randomized in a 2:1 ratio to receive either efgartigimod IV or placebo IV. At the end of the treatment period (up to 24 weeks), all participants will receive efgartigimod IV during the first year open-label treatment period (OLTP1). At the end of the first OLTP1, participants may begin a second year (OLTP2). After the OLTP2, the participants will enter a follow-up period (approximately 8 weeks) while off study drug. The participants will be in the study for up to 138 weeks

ELIGIBILITY:
Inclusion Criteria:

* Is aged 12 to less than 18 years when completing the informed consent process
* Has a documented duration of primary ITP of more than 12 months on the date the informed consent process is complete
* Has documented prior ITP treatment with at least 1 of the following treatments: corticosteroids, IVIg, anti-D immunoglobulin, thrombopoietin receptor agonist (TPO-RAs), or rituximab.
* Has documented prior response, defined as 1 platelet count of ≥50 × 10^9/L to at least 1 of the following ITP treatments: prednisone, other or nonspecified corticosteroids, IVIg, or anti-D immunoglobulin
* Has documented insufficient response to a prior ITP treatment with corticosteroids, IVIg, anti-D immunoglobulin, TPO-RAs, rituximab, or splenectomy
* Has documented mean platelet count of less than 30 x10^9/L

Exclusion Criteria:

* Secondary ITP according to the following definition by the International Working Group (IWG): all forms of immune-mediated thrombocytopenia except primary ITP
* Nonimmune thrombocytopenia
* ITP-associated critical or severe bleeding
* History of hereditary thrombocytopenia

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Efgartigimod serum concentrations in the DBTP | Up to 24 weeks
Total IgG levels in the DBTP | Up to 24 weeks

SECONDARY OUTCOMES:
Efgartigimod serum concentrations over time during the DBTP | Up to 24 weeks
Percent change from baseline in total IgG levels in serum over time during the DBTP | Up to 24 weeks
Incidence of AEs, SAEs and AEs leading to IMP discontinuation | Up to 136 weeks
  SAE: Serious adverse event; AE: adverse event
Sustained platelet count response between study weeks 19 and 24 of the DBTP and in OLTP1 for participants receiving placebo in the DBTP | Up to 48 weeks
  Sustained platelet count defined as achieving platelet counts of ≥50 × 10^9/L for at least 4 of the 6 study visits
Extent of disease control during the DBTP and during the first 24 weeks of OLTP1 for those participants receiving placebo in the DBTP | Up to 48 weeks
  Extend of disease defined as the number of cumulative weeks with a platelet count of ≥50 × 10^9/L
Changes from baseline for platelet counts over time | Up to 76 weeks
Incidence of bleeding, assessed by the Modified Buchanan and Adix Bleeding Score for pediatric ITP | Up to 76 weeks
  The Modified Buchanan and Adix Bleeding Score for pediatric ITP is a semiquantitative assessment tool that measures bleeding signs and symptoms, comprising a score based on a scale of 0 to 5, each representing a different level of severity (0 = no risk; 5 = highest severity).
Incidence of ADA and Nab against efgartigimod in serum | Up to 76 weeks
  ADA: anti-drug antibodies; Nab: neutralizing antibodies
Change from baseline in EQ-5D-5L | Up to 76 weeks
  The European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) is a questionnaire comprised of 5 dimensions. Participants are asked to select the statement in each dimension which best describes their health on the day they complete the questionnaire. Responses in each dimension are coded as a 1-digit number ranging from 1 (no problems) to 5 (extreme problems).
Change from baseline in KIT Child Self-Report and KIT Parent Impact Report | Up to 76 weeks
  The Kids' ITP Tools (KIT) comprises two disease- specific tools: a self-report form for children aged 12 and older, and a parent impact form. Respondents provide insights into their disease experience using a 1-week recall period. The instrument generates a total score, calculated by summing the items and converting them to a scale of 0 to 100, where higher scores reflect a better disease-specific quality of life (QoL).
Change from baseline in peds FACIT-F | Up to 76 weeks
  In all participants, the pediatric Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) will use to assess health-related quality of life (HRQoL) before and after treatment. The FACIT-F questionnaire has a score range of 0 to 52, where 0 represents the worst possible fatigue and 52 indicates no fatigue.

CONTACTS AND LOCATIONS:
Locations (7):
- Uniwersytecki Szpital Dzieciecy w Lublinie, Lublin, Poland
- Institutul Clinic Fundeni, Bucharest, Romania
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Deu Barcelona, Esplugues de Llobregat
  - Hospital Infantil Universitario Nino Jesus (HIUNJS), Madrid
  - Hospital Materno-Infantil Universitario Gregorio Maranon, Madrid
- Cardiff and Vale NHS Trust - University Hospital of Wales (UHW), Cardiff, United Kingdom

IPD SHARING:
Plan to Share IPD: No